CLINICAL TRIAL: NCT05201677
Title: Improved Operation of Low Intraocular Pressure in Phacoemulsification for Patients With High Myopia Complicated With Cataract
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yune Zhao (Other)
Responsible Party: Sponsor-Investigator, Yune Zhao, Vice president of Eye Hospital of Wenzhou Medical University, Wenzhou Medical University
Organization: Wenzhou Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WDD-High myopia-Low IOP
Record Dates: First submitted 2021-11-23; First posted 2022-01-21 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: High Myopia; Low Intraocular Pressure
MeSH Terms: conditions — Ocular Hypotension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High myopia with axial length between 26 mm and 28 mm (Experimental): The patients' axial length is between 26 mm and 28 mm
  Interventions: Procedure: Supplement of perfusion fluid through the subiris suspensory ligament space from the lateral incision
- High myopia with axial length more than 28 mm (Experimental): The patients' axial length is more than 28 mm
  Interventions: Procedure: Supplement of perfusion fluid through the subiris suspensory ligament space from the lateral incision

INTERVENTIONS:
Procedure: Supplement of perfusion fluid through the subiris suspensory ligament space from the lateral incision — After the capsule is filled with viscoelastic material, if the IOP is less than 10 mmHg, the investigators will supply the perfusion fluid through the subiris suspensory ligament space from the lateral incision.

SUMMARY:
Approximately 60 participants at Eye Hospital of Wenzhou Medical University during October,2021 to January 2022 will be enroll in the investigators' study. And dived them randomly into 2 groups:High myopia with axial length between 26 mm and 28 mm and High myopia with axial length more than 28 mm (30 eyes) .

ELIGIBILITY:
Inclusion Criteria:

* The patients with high myopia and cataract who plan to receive cataract surgery in our hospital
* Surgery without complications

Exclusion Criteria:

* Patients who had other ocular diseases or had undergone internal eye surgery
* Patients with a history of myopic laser surgery
* Previous history of eye trauma
* Previous use of medications/eye drops that may alter IOP

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Intraocular pressure | two minutes
  Measurement of intraocular pressure during cataract surgery by iCare rebound tonometer

CONTACTS AND LOCATIONS:
Locations (1):
- Eye Hospital of Wenzhou Medical College, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wang D, Shi J, Guan W, Zhu M, Lou X, Zhao Y, Chang P, Zhao Y. Fluid Supplementation Through Weakened Zonules via Side-Port Incision to Maintain Intraocular Pressure in High Myopic Eyes. Ophthalmol Ther. 2023 Dec;12(6):3323-3336. doi: 10.1007/s40123-023-00814-w. Epub 2023 Oct 9. PMID 37812307